CLINICAL TRIAL: NCT02776943
Title: Phase I/II Study of Umbilical Cord Mesenchymal Stem Cell Implantation in the Treatment of Articular Cartilage Defect of Knee and Knee Osteoarthritis
Brief Title: UCMSC Transplantation in the Treatment of Cartilage Damage
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South China Research Center for Stem Cell and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCMSC-4
Record Dates: First submitted 2016-03-14; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-01

CONDITIONS: Cartilage Damage; Degenerative Osteoarthritis
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cell treatment (Experimental): Umbilical Cord Mesenchymal stem cells (UCMSC) expanded and treated for 1-2 weeks. Then administer 5x10^6 of UCMSC per cm^2 of the cartilage defect.
  Interventions: Biological: umbilical cord mesenchymal stem cells
- Hyaluronic acid treatment (Active Comparator): Administer hyaluronic acid (30 mg) in a single injection
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells
  Other Names: UCMSC
  Arms: Mesenchymal stem cell treatment
Device: Hyaluronic acid
  Arms: Hyaluronic acid treatment

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of transplantation of umbilical cord mesenchymal stem cells（UCMSCs） in patient with Knee cartilage damage.

DETAILED DESCRIPTION:
Human cartilage only has limited regenerative potential. Transplantation of umbilical cord mesenchymal stem cells (UCMSCs) is a promising strategy given the high proliferative capacity of MSCs and their potential to differentiate into cartilage-producing cells - chondrocytes. The acquisition of ucMSCs does not require invasive surgical intervention or cartilage extraction from other sites as required by other cell-based strategies. The investigators inject allogeneic human mesenchymal stem cells to the cartilage lesions in patients via intra-articular injection method, and to investigate the efficacy and safety。

ELIGIBILITY:
Inclusion Criteria:

* Patients whose lesion (single joint) should be in the range of 2 cm^2-8 cm^2.
* Patients with pain in affected joint of 60 mm- 100 mm VAS (visual analogue scale)
* Patients with articular swelling, tenderness and active range of motion of Grade 2 or below
* Patients with knee joint cartilage defect or injury of ICRS (International Cartilage Repair Society) Grade 4 confirmed by arthroscopy (At screening, patients diagnosed as such with an MRI may be included)
* Patients who needs invasive interventions of arthroplasty due to no response from existing pain medication
* Patients voluntarily agreed to participate in the study and signed informed consent

Exclusion Criteria:

* Patients with autoimmune diseases or medical history
* Patients with infections requiring injection of antibiotics
* Patients with severe internal diseases
* Patients who are currently pregnant or lactation
* Patients who had participated in any other clinical trials within the past four weeks
* Patients who had been administered with immunosuppressants within the past four weeks
* Patients whom the principal investigator considers inappropriate for the clinical trial due to any other reasons than those listed above

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Knee Function Change and Improvement | 12 months after treatment
  Knee assessments will be performed using the following tools:
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Knee Function Change and Improvement | 12 months after treatment
  Changes in knee function will be assessed via the IKDC score.

SECONDARY OUTCOMES:
Severity of adverse events | 12 months
  Adverse events were categorized using National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.0 scale (NCI-CTCAE v4.0)

IPD SHARING:
Plan to Share IPD: No